CLINICAL TRIAL: NCT04736992
Title: HKCFP-HKU Primary Care Morbidity Survey in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Julie Yun Chen, Associate Professor (Teaching), The University of Hong Kong
Other Study IDs: HKUCTR-2916
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Primary Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention involved — No intervention involved

SUMMARY:
Background:

Information about the health problems of patients presenting in primary care is crucial to understanding the health of the general community for the planning and allocation of health care resources. Practice-based morbidity studies conducted in primary care settings have proven to be helpful in documentation of disease prevalence and for service planning. With the change in morbidity pattern and the aging population, our study will help to inform primary health care policy and guide work force and service planning.

Method:

This is a prospective practice-based study of health problems presenting in primary care. Doctors who agree to participate in the study will record the health problem and type of management performed in consecutive patient encounters for one of the designated weeks during each season over the course of one year.

Analysis:

Data collected will be analysed by descriptive statistics, comparison with data from previous morbidity study, and by non-linear mixed effects for factors associated with morbidity and management patterns in primary care.

Results:

Findings will will 1) provide evidence to support the allocation of resources to continue and to expand primary care initiatives that support the provision of quality chronic disease care in private sector, 2) enable continued surveillance of the morbidity trends in Hong Kong by providing data for comparison with past and future studies, and 3) inform the content of educational curricula for medical and health care students and practitioners to prepare them to better meet the needs of the community.

ELIGIBILITY:
Inclusion Criteria:

* Consented primary care doctors in Hong Kong who are working in:
* the public sector (GOPC), or
* Department of Health Clinic, or
* private solo or group practices, or
* university health services, or
* non-profit organizations, or
* private hospital family medicine clinics

Exclusion Criteria:

* Doctors who do not consent
* Doctors who are not working as primary care doctors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care doctors in Hong Kong who are working in the public sector (GOPC), Department of Health Clinic, private solo practices, university health services, non-profit organizations and private hospital family medicine clinics
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of health problems and diseases presenting in primary care | immediately after completion of data collection, up to 6 months
Rates of management activities including referral, investigation, prescription and preventive care intervention by primary care doctors | immediately after completion of data collection, up to 6 months
Distribution of health problems and diseases presenting in the public compared with the private primary care setting | immediately after completion of data collection, up to 6 months
Factors which affect the proportion and distribution of health problems in the public sector compared with the private sector | immediately after completion of data collection, up to 6 months

SECONDARY OUTCOMES:
Prescription rates of specific classes of drugs including benzodiazepines, antidepressants, NSAIDs, and antibiotics | immediately after completion of data collection, up to 6 months
Seasonal variation in primary care morbidity pattern | immediately after completion of data collection, up to 6 months
Relationship between patient's presenting problem and doctor's diagnosis | immediately after completion of data collection, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Y Chen, MD, Principal Investigator — Department of Family Medicine and Primary Care, University of Hong Kong; Cindy LK Lam, MD, Principal Investigator — Department of Family Medicine and Primary Care, University of Hong Kong
Locations (1):
- Department of Family Medicine and Primary Care, University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Chen JY, Chao D, Wong SY, Tse TYE, Wan EYF, Tsang JPY, Leung MKW, Ko W, Li YC, Chen C, Luk W, Dao MC, Wong M, Leung WM, Lam CLK. Morbidity Patterns in Primary Care in Hong Kong: Protocol for a Practice-Based Morbidity Survey. JMIR Res Protoc. 2022 Jun 22;11(6):e37334. doi: 10.2196/37334. PMID 35731566